CLINICAL TRIAL: NCT02007798
Title: Randomized, Parallelled and Double-blinded Trial of Small-dose Dexmedetomidine Effects on Recovery Profiles of Supratentorial Tumors Patients From General Anesthesia
Brief Title: Small-dose Dexmedetomidine Effects on Recovery Profiles of Supratentorial Tumors Patients From General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yue Yun, Randomized, parallelled and double-blinded trial of small-dose dexmedetomidine effects on recovery profiles of supratentorial tumors patients from general anesthesia, China Medical University, China
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CMU-1st-001
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Brain Neoplasms; Surgery
Keywords: dexmedetomidine; supratentorial tumors
MeSH Terms: conditions — Brain Neoplasms; Supratentorial Neoplasms | interventions — Dexmedetomidine; Long-Term Synaptic Depression; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low-dose group (Experimental): S group : dexmedetomidine is infused intravenously at a dose of 0.4 ug/kg
  Interventions: Drug: dexmedetomidine
- middle-dose group (Experimental): M group: dexmedetomidine is infused intravenously at a dose of 0.8 ug/kg
  Interventions: Drug: dexmedetomidine
- control group (Experimental): P group: normal saline is infused intravenously
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: dexmedetomidine — 2 ml of dexmedetomidine at a concentration of 100 ug/ml is diluted by 98 ml normal saline to a concentration of 2 ug/ml. The required amount of experimental drugs is confirmed according to the weight and grouping, and diluted using normal saline to 20 ml.
  Other Names: SFDA Approval No. H20090248; produced by Jiangsu Hengrui Medicine Co., Ltd., China.
  Arms: low-dose group; middle-dose group
Drug: normal saline — 100 ml per bag
  Other Names: provided by the Central Pharmacy of the hospital
  Arms: control group

SUMMARY:
An excellent recovery profile is critical for neurosurgical anesthesia. Rapid awakening, smooth blood pressure and heart rate (HR), a higher degree of coordination, painless or mild pain, as well as better tolerance to endotracheal intubation can avoid can increased intracranial pressure, elevated blood pressure and rapid HR caused by emergency choking, suffocation and agitation, and can reduce postoperative cerebral edema and the risk of bleeding. In addition, it is easy for surgeons to timely evaluate postoperative patients' neurologic function based on the excellent recovery from anesthesia. Up to now, there are many methods and drugs to improve the quality of recovery period, but each of them has some flaws. Dexmedetomidine, an emerging anesthetic adjuvant, exhibits a stable hemodynamic recovery period, and cannot affect evaluation of neurological function with both the sedative and analgesic effects. We propose the following hypotheses: (1) A small dose of dexmedetomidine can be intravenously injected into patients subjected to craniotomy under general anesthesia, in order to improve the recovery profiles and reduce the incidence of emergence agitation. (2) Dexmedetomidine can reduce postoperative pain.

DETAILED DESCRIPTION:
Study Arm(s):

Enrollment There are totally 150 cases, 50 cases in each group. At least 120 cases complete the test.

Randomized grouping Under the guidance of a drug administrator, the different drug and control groups are randomly encoded. Each code has a corresponding emergency envelope. Blind codes are saved by the drug administrator.

Interventions :

Experimental Drugs Dexmedetomidine (SFDA Approval No. H20090248), 200 ug/2 ml, provided by the Central Pharmacy of the First Affiliated Hospital of China Medical University and produced by Jiangsu Hengrui Medicine Co., Ltd., China.

Normal saline, 100 ml per bag, provided by the the Central Pharmacy of the First Affiliated Hospital of China Medical University.

Experimental Procedures:

Background Information: Dexmedetomidine is an α-adrenoceptor agonist, and its chemical name is (+)-4-(S)-[1-(2,3-dimethylphenyl ) ethyl]-1H-imidazole hydrochloride. Its structure and pharmacological activity are similar to clonidine. Dexmedetomidine was developed by the Orion Pharma (Finland) Corporation and Abott (USA), and introduced to China in 2009 (trade name: Ai Beining). Preclinical studies have shown that, like clonidine, dexmedetomidine is an agonist of α2-adrenergic receptors, and exhibits effectiveness about 10 times more than clonidine. Originally developed as an antihypertensive drug, dexmedetomidine functions in lowering blood pressure and HR, and is found to have a powerful anesthetic effect. Up to now, dexmedetomidine has been widely used in general anesthesia, monitored anesthesia care (MAC), ICU sedation. Dexmedetomidine is a sedative, hypnotic, analgesic, anti-sympathetic medication, and uniquely characterized as "cooperative sedation" and "no respiratory depression".

In the present study, we compare the hemodynamic effects of different doses of dexmedetomidine via intraoperative infusion, and explore the effects of dexmedetomidine on recovery profiles from general anesthesia and postoperative pain.

Experimental Protocol:

This study is a randomized double-blinded trial. All the subjects are supratentorial brain tumors patients with ASA I & II. Within 24 hours before surgery, preoperative visits are conducted to obtain signed informed consents. The patient's height, weight, blood pressure (including SBP, DBP and mean arterial pressure (MAP)), HR, oxygen saturation (SpO2) are recorded as the baseline value (BV).

Patients are subjected to electrocardiograph monitoring, including non-invasive blood pressure, ECG, and SpO2.

Anesthesia is orderly induced by a combined infusion of propofol 2-2.5 mg/kg, sufentanil 0.3-0.5 ug/kg, and cis-atracurium 0.15-0.2 mg/kg, and the tracheal intubation is completed until the maximal muscle relaxant effect.

Before surgery, arterial and central venous catheterization is completed for continuous monitoring of the patient's arterial pressure and central venous pressure (CVP). Intraoperative CVP is maintained at 4-6 cmH2O.

Anesthesia is maintained at a manner of inhalation anesthesia with 0.8-1.5% sevoflurane and continuous intravenous infusion of propofol and remifentanil respectively at a speed of 3-5 mg/kg/h and 0.01-0.02 mg /kg/h. The drug dose is adjusted hemodynamically to maintain MAP values at a range of 60-90 mmHg.

After craniectomy, additional cis-atracurium 0.05-0.08 mg/kg is added every 45-60 minutes by the end of dural suturing. Sufentanil (0.15-0.2 ug/kg) is given intravenously instead of inhalation anesthesia, and meanwhile, 20% -30% dose of intravenous anesthesia is added. After skin closure (approximately 30 minutes before the end of surgery), continuous infusion of propofol is terminated, and remifentanil infusion is stopped after surgery. Intraoperative dexamethasone (20 mg) is routinely used for prevention of cerebral edema, 10 mg is administered intravenously before surgery (10 mg), and then an additional 10 mg injected after 2 hours or by the end of surgery.

Infusion principles: before anesthesia, crystalloid solution is dropped at a speed of 8-10 ml/kg/h. After the start of anesthesia, the infusion speed is adjusted to 5ml/kg/h. The dose of artificial colloids is less than 20 ml/kg. The infusion volume is adjusted based on the amount of fluid input and output.

Experimental drugs are infused via the syringe pump approximately 1 hour before the end of surgery, i.e., at the end of dural suturing, at a speed of 2 ml/min, i.e., 120 ml/h.

Criteria for extubation: a. recovery of spontaneous breathing; b. over 95% SpO2; c. patients can complete the instructions (eye opening to voice).

Criteria for discharge from the Post Anesthesia Care Unit (PACU): a. 1<= RASS score> = -2; b. in the case of oxygen inhalation via a nasal catheter at a flow rate of 3-5 L/min, SpO2 can maintain above 95%; c. the observation time after extubation is > = 30 minutes.

Medical equipments used in surgery: GE healthcare SolarTM8000M/i Patient Monitor; GE healthcare Smart Anesthesia Multi-gas SAMTM/SAM-80 Module (multi-gas analyzer); Drager Fabius GS; JMS syringe pump (SP-500).

Medical equipments used in PACU: GE healthcare B30 Patient Monitor; NHI ventilator (Newport Medical Instruments, Inc., USA).

Medical equipments used in Neurosurgical intensive care unit (NICU): GE Dash 2500 Monitor; GEM Premier 3000 blood gas analyzer.

Adverse Events:

All the adverse events occur after drug administration, which may be unrelated to drug treatment.

Observation and recording of adverse effects Careful inquiry and tracing is necessary for all the adverse events during the experiment, including laboratory abnormalities. All adverse events must be judged by their nature, severity and correlation with drug treatment, which should be strictly recorded in the case report form.

Correlation assessment Correlations between adverse events and experimental medication are as follows: definitely related, probably related, possibly related, possibly unrelated, certainly unrelated. The incidence of adverse reactions is calculated based on three conditions described as definitely related, probably related, and possibly related. Specific criteria are seen in Appendix 1.

Severity assessment

Severity of adverse events is divided into three levels:

Mild: Treatment is usually not necessary for a transient increase in blood pressure and decrease in HR, because the subject is under anesthesia.

Moderate: The bolus injection of atropine 0.3-1 mg is given for sinus bradycardia and escape rhythm. If combination with hypotension, the bolus injection of ephedrine 10-15 mg can be applied.

Severe: For sinus standstill, cardiopulmonary resuscitation is applied if necessary.

Treatment for adverse events during and after the experiment Outcomes of all adverse events should be followed and recorded. The subject who withdraws from the experiment due to adverse events should be traced till the adverse events completed removed. Researchers must determine whether an adverse event is related to experimental drugs, and provide a basis to support this judgment.

Serious adverse events Definition: Adverse events occur during clinical trials that result in a series of serious consequences, including hospitalization, prolonging hospitalization, disability, affecting the ability to work, endangering the life or death, and congenital malformations.

Reporting of the serious adverse events: Serious adverse reactions should be reported to the team leader and sponsor within 24 hours, and the serious adverse event table should be filled.

Contacts: Yue Yun, +86 13889168717, Second Department of Anesthesiology First Affiliated Hospital of China Medical University, China Urgent Unblinding Method When serious adverse reactions appear during the experiment, if necessary, the study director can open the emergency envelope to carry out urgent unblinding strategy and record the relevant causes and date in the case report form. Whether the unblinded subjects withdraw from the experiment is decided by investigators and responsible party.

Data management and Statistical Analyses:

Statistical Description: Completed case report forms are collected by the clinical inspector and submitted to the responsible party for data processing.

After confirmation, the data from case report forms are locked into the database.

There are 3 groups when unblinding for the first time. Information description Count data are described using percentages, and measurement data expressed as mean ± standard deviation. Not normally distributed data are expressed as median and percentiles (25th-75th percentiles).

Comparison of baseline data Intergroup count data are compared using chi-square test or Fisher's exact test. If measurement data normally distributed exhibit homogeneity of variance, single-factor or multi-factor analysis of variance is applied. If heterogeneity of variance is shown, non-parametric test or approximate test (e.g., Tamhnnes T2 test) is employed. For measurement data not normally distributed, non-parametric Mann-Whitney U test or Kruskall-Wallis rank sum test is used. Baseline balance and comparability in each group is examined.

Comparison of Efficacy: Analgesic and sedative effects between groups are compared using Kruskall-Wallis rank sum test. For markedly effective, pairwise comparison in data differences between are analyzed using Mann-Whitney U non-parametric test. Considering the center or other factors, CMH X2 test is employed for comparison of two-classification index and level indicators.

Data Processing: All statistical data are analyzed using SAS software for data processing. Two-sided test is employed for statistical analysis, and the corresponding P values are given. For the Fisher's exact test, P value is calculated directly. A value of P <0.05 is considered significant, and P <0.01 considered highly significant.

Unblinding for the second time is carried out by the end of statistical analysis, and there are two experimental groups and one control group.

Quality Assurance and Quality Control:

Investigators In this clinical study, there are two responsible parties and five principal investigators. The clinical scheme is implemented strictly. An inspector is appointed to monitor the clinical trial at any time.

Quality Control of the measurement indexes The observation indexes are observed according to standard operating procedures and quality control procedures. National legal units of measurements are employed for various test items. The test report form must complete the Assay report card must have complete items, including the date, test items, test results and their normal range.

Ethical standards The study protocol, case report forms, informed consent should be approved by the Ethics Committee of the First Affiliated Hospital of China Medical University.

Investigators or investigator-authorized officers will be responsible to explain the benefits and risks of participating in the clinical trial for each patient, the patient's legal representative or notary witnesses. The written informed consent should be obtained prior to study entry (before screening test and drug administration).

All the patients or their legal representatives and personnel chairing the informed consent process sign their names and date to the informed consent. The original file is saved by the investigators.

Data retention The investigators should be responsible for the intact data intact, have a fixed place to store the data which are locked for future viewing. In accordance with the principles of GCP in China, the data should be kept for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist class (ASA) I & II (ASA I: normal healthy patient; ASA II: patient with mild systemic disease; no functional limitation)；Preoperative MRI diagnosis of supratentorial lesions (glioma, meningioma or neurofibroma), and tumor diameter <= 40 mm；The subject gets full score for Glasgow Coma Score；Estimated operation time <= 6 hours and anesthesia time <= 8 hours；The subject has given written informed consent.

Exclusion Criteria:

* The subject has participated in other clinical trials at 4 weeks before the beginning of the present study；The subject is taking or has taken β-blockers (such as metoprolol) within 2 weeks before the beginning of the present study；The subject has undergone craniotomy twice or more；The subject has a history of sinus bradycardia (preoperative electrocardiogram of HR <= 50 beats/min), sick sinus syndrome, myocardial infarction, Ⅱ grade and grade Ⅱ cardiac function, and severe hypertension (systolic blood pressure (SBP)> = 180 mmHg or diastolic blood pressure (DBP)> = 110 mmHg)；The subject has a history of lung disease (blood oxygen content <95% when breathing air at an awake state)；The subject has a history of liver dysfunction (1.5 times or more that of the normal value)；The subject has a history of kidney dysfunction (levels of serum creatinine and blood urea nitrogen are out of the normal range)；Hypersensitivity to dexmedetomidine；Tolerance to dexmedetomidine；The subject has a history of drugs or alcohol abuse；The weight exceeds ±15% of standard weight range, and the standard weight is calculated as the following formula: standard weight=body height (cm)-100；Pregnant or lactating women；The subject is considered unsuitable for this trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic impacts | Up to 240 minutes after returning to the ward
  Patients' SBP, DBP, MAP and HR are recorded before and every 5 minutes after drug intervention until recovery from anesthesia and removal of the tracheal intubation.
  Record SBP, DBP, MAP, HR, and SpO2 values immediately after extubation. Record SBP, DBP, MAP, HR, and SpO2 values every 5 minutes after extubation. Record SBP, DBP, MAP, HR, and SpO2 values every 5 minutes after PACU entry. Record SBP, DBP, MAP, HR, and SpO2 values at 0, 60, 120 and 240 minutes after returning to the ward.

SECONDARY OUTCOMES:
Time of recovery from anesthesia | From the anesthetic induction to extubation
  Record the patient's anesthesia time (from the anesthetic induction to termination of anesthetic infusion), operative time (from skin incision to the end of suturing), awakening time (from the end of surgery to eye opening in response to voices), spontaneous breathing recovery time (from the end of surgery to recovery of spontaneous breathing), extubation time (from the end of surgery to extubation).
Cough assessment at tracheal extubation | At tracheal extubation
  Using Four-point subjective scale: 0 = no cough; 1 = mild cough; 2 = moderate cough; 3 = severe cough.
Degree of sedation | At tracheal extubation, every 5 minutes after extubation, and at 0, 30, 60, 120, 240 minutes after returning to the ward
  Richmond Agitation-Sedation Scale (RASS) is used for sedation assessment. Scores on RASS are recorded at tracheal extubation, every 5 minutes after extubation, and at 0, 30, 60, 120, 240 minutes after returning to the ward.
  If RASS>=2 during emergence from general anesthesia, the bolus injection of propofol 1.5-2.5mg/kg can be applied when necessary.
Sedative effectiveness | Up to 240 minutes after returning to the ward
  Verbal numerical rating scale (VNRS) is employed for assessment of pain intensity (PI). The scores range from 0-10: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, and 7-10 = severe pain.
  In the operation room, the subject is asked to say the VNRS scores by the PACU nurse, and the score is recorded. The VNRS assessment is also conducted at 5, 15, 30 minutes after recovery from anesthesia, and at 0, 30, 60, 120, 240 minutes after returning to the ward.
  During emergence from general anesthesia, if VNRS score> = 6 points, a single-dose bolus injection of sufentanil 5 ug is applied; if pain is not alleviated, sufentanil 5 ug can be given again after 5 minutes, and total dose does not exceed 10 ug.
Test patient's blood pressure during maintenance of anesthesia | During maintenance of anesthesia
  When MAP> 90 mmHg during maintenance of anesthesia, the amount of anesthetic drugs will be increased, i.e. the inhalation concentration of sevoflurane, propofol and/or remifentanil infusion dose. If the result is still not satisfactory, a single dose of nicardipine 0.5-1 mg via intravenous injection will be added.
  When MAP <60 mmHg, a single intravenous injection of ephedrine 5-10 mg can be given, while the value of MAP also can be adjusted by fluid replacement and reducing anesthetic doses (such as the inhalation concentration of sevoflurane, propofol, and/or remifentanil infusion dose) to adjust; if the effect is still not satisfactory, continuous infusion of 2% norepinephrine is recommended to maintain blood pressure in the target range.
Monitor Patient's heart beat during maintenance of anesthesia | During maintenance of anesthesia
  When HR> 90 beats/min or ST-T segment abnormalities on ECG appear during maintenance of anesthesia, a single dose of 5-10 mg esmolol can be given intravenously, and meanwhile, the fluid replacement is recommended. When HR <45 beats/min, a single dose of 0.3-0.5 mg atropine can be given intravenously; if the result is not satisfactory and repeated administration is up to the maximum cumulative amount of 2 mg, isoproterenol 1 mg/500 ml can be given intravenously and the infusion speed can be adjusted based on HR.
Test patient's blood pressure during anesthesia recovery period | During anesthesia recovery period
  If MAP> BV +20% lasts more than 1 minute during anesthesia recovery period, a single-dose bolus injection of nicardipine 0.5-1mg is given; if the result is not satisfactory, repeated doses (nicardipine 10 mg/100 ml) and the infusion rate can be adjusted according to blood pressure values.
  If MAP <70 mmHg lasts more than 1 minute, a single-dose bolus injection of ephedrine 5-10 mg bolus is preferred, and meanwhile, the fluid replacement is also introduced under the premise of exclusion of cardiogenic shock; if necessary, continuous infusion of 2% norepinephrine can be given to maintain the blood pressure in the target range.
Monitor Patient's heart beat during anesthesia recovery period | during anesthesia recovery period
  When HR> 120 beats/min or ST-T segment abnormalities on ECG appear during anesthesia recovery period, a load dose of esmolol 5-10 mg is necessary followed by continuous intravenous infusion of esmolol 100 mg/100 ml to control HR. The infusion rate is adjusted according to the value of HR.
  When HR <45 beats/min, the bolus injection of atropine 0.3-0.5 mg is given; if the result is not satisfactory and repeated administration is up to the maximum cumulative amount of 2 mg, repeated administration to the maximum cumulative amount 2mg, the intravenous infusion of isoproterenol 1 mg/500 ml can be given and the infusion rate is adjusted according to the HR value.
Observe chills reaction | At emerge from general anesthesia
  If chills reaction appear when the patient emerges from general anesthesia, the intravenous injection of tramadol hydrochloride 0.1 g should be given slowly on the basis of heat preservation; if appearance of nausea and vomiting, the intravenous injection of tropisetron hydrochloride (Xinbei) 5 mg should be given.
To measure palinesthesia | At emerge from general anesthesia
  Palinesthesia is evaluated by the surgeon based on a visual analogue scale VAS 0-10 points: 0=dissatisfied, 10=very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Pei, Principal Investigator — Department of Anesthesiology, the First Affiliated Hospital of China Medical University, China
Locations (1):
- Yue Yun, Shenyang, Liaoning, China